CLINICAL TRIAL: NCT01313299
Title: A Phase III, Multicentre, Prospective, Double Blind, Randomised, Placebo Controlled Study, Assessing the Efficacy and Safety of Dysport® Intramuscular Injections Used for the Treatment of Upper Limb Spasticity in Adult Subjects With Spastic Hemiparesis Due to Stroke or Traumatic Brain Injury
Brief Title: Dysport® Adult Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y-52-52120-145; 2010-019069-28 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Nervous System Disorders
MeSH Terms: conditions — Nervous System Diseases | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Dysport 500 U (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Dysport 1000 U (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — 500 U, I.M. (in the muscle) injection on day 1 of a single treatment cycle.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport 500 U
Biological: Botulinum toxin type A — 1000 U, I.M. (in the muscle) injection on day 1 of a single treatment cycle.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport 1000 U
Drug: Placebo — I.M. (in the muscle) injection on day 1 of a single treatment cycle.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to assess the efficacy of Dysport compared to placebo in improving muscle tone in hemiparetic subjects with upper limb spasticity due to stroke or traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients - post stroke or brain injury
* Modified Ashworth Scale ≥ 2
* Ambulatory patients

Exclusion Criteria:

* Previous treatment with botulinum toxin of any type within 4 months prior to study entry for any condition
* Physiotherapy initiated less than 4 weeks before inclusion
* Previous surgery, alcohol, phenol in upper limb
* Neurological/neuromuscular disorders which may interfere with protocol evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (40):
- United States (15):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Associated Neurologist of Southern CT, PT, Fairfield, Connecticut
  - Parkinson's Disease & Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Design Neuroscience Miami, South Miami, Florida
  - The Rehabilitation Institute of Chicago, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Univ of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, Dallas, Texas
  - Southwestern Medical Center at Dallas, Dallas, Texas
  - University of North Texas HSC, Fort Worth, Texas
  - University of Texas, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Belgium (2):
  - Université catholique de Louvain av Hippocrate 10, Brussels
  - Clinique Universitaire, Yvoir
- Czechia (2):
  - Neurologicka klinika, Olomouc, Olomouc
  - Charles University in Prague, Prague
- France (8):
  - CHU Jean MINJOZ, Besançon
  - CHU Brest, Brest
  - Centre de Réadaptation de Coubert, Coubert
  - Centre Hospitalier Albert Chenevier-Hopital Henri Mondor, Créteil
  - Hopital Raymond Poincarré, Garches
  - Hôpital Sébastopol, Reims
  - CHU Strasbourg, Strasbourg
  - Hopital Rangueil, Toulouse
- Hungary (3):
  - National Institut for Medical Rehabilitation, Budapest
  - Petz Aladar County Hospital, Győr
  - University of Szeged, Szeged
- Italy (2):
  - Azienda Hospedaliero, Catania
  - Policlinico Universitario Agostino Gemelli, Roma
- Poland (3):
  - Malopolskie Centrum Medyczne, Krakow
  - Krakowska Akademia Neurologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Russia (3):
  - Medical Rehabilitation Center, Moscow
  - Scientific Center of Neurology of RAMS, Moscow
  - State University, Saint Petersburg
- Slovakia (2):
  - Derer's Hospital, Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Delafont B, Carroll K, Vilain C, Pham E. Investigation of mixed model repeated measures analyses and non-linear random coefficient models in the context of long-term efficacy data. Pharm Stat. 2018 Sep;17(5):515-526. doi: 10.1002/pst.1868. Epub 2018 May 20. PMID 29781237
- [Derived] O'Dell MW, Brashear A, Jech R, Lejeune T, Marque P, Bensmail D, Ayyoub Z, Simpson DM, Volteau M, Vilain C, Picaut P, Gracies JM. Dose-Dependent Effects of AbobotulinumtoxinA (Dysport) on Spasticity and Active Movements in Adults With Upper Limb Spasticity: Secondary Analysis of a Phase 3 Study. PM R. 2018 Jan;10(1):1-10. doi: 10.1016/j.pmrj.2017.06.008. Epub 2017 Jun 19. PMID 28634000
- [Derived] Marciniak C, McAllister P, Walker H, Brashear A, Edgley S, Deltombe T, Khatkova S, Banach M, Gul F, Vilain C, Picaut P, Grandoulier AS, Gracies JM; International AbobotulinumtoxinA Adult Upper Limb Spasticity Study Group. Efficacy and Safety of AbobotulinumtoxinA (Dysport) for the Treatment of Hemiparesis in Adults With Upper Limb Spasticity Previously Treated With Botulinum Toxin: Subanalysis From a Phase 3 Randomized Controlled Trial. PM R. 2017 Dec;9(12):1181-1190. doi: 10.1016/j.pmrj.2017.06.007. Epub 2017 Jun 16. PMID 28625615
- [Derived] Gracies JM, Brashear A, Jech R, McAllister P, Banach M, Valkovic P, Walker H, Marciniak C, Deltombe T, Skoromets A, Khatkova S, Edgley S, Gul F, Catus F, De Fer BB, Vilain C, Picaut P; International AbobotulinumtoxinA Adult Upper Limb Spasticity Study Group. Safety and efficacy of abobotulinumtoxinA for hemiparesis in adults with upper limb spasticity after stroke or traumatic brain injury: a double-blind randomised controlled trial. Lancet Neurol. 2015 Oct;14(10):992-1001. doi: 10.1016/S1474-4422(15)00216-1. Epub 2015 Aug 26. PMID 26318836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in 34 investigational sites. Subjects screened were 281 and randomised and treated were 243.
Groups:
- Placebo: Placebo intramuscular injection single treatment cycle on day 1
- Dysport 500 U: Botulinum type A toxin (Dysport) 500 U intramuscular injection single treatment cycle on day 1
- Dysport 1000 U: Botulinum type A toxin (Dysport) 1000 U intramuscular injection single treatment cycle on day 1
Period: Overall Study
Arm/Group | Placebo | Dysport 500 U | Dysport 1000 U
Started | 81 | 81 | 81
Completed | 74 | 78 | 77
Not Completed | 7 | 3 | 4
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Family reason and moved out of state | 0 | 2 | 0
Not completed — Lack of subject compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport 500 U | Dysport 1000 U | Total
Number analyzed (Participants) | 81 | 81 | 81 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.8) | 52.8 (12.8) | 53.2 (13.8) | 52.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 28 | 87
  Male | 50 | 53 | 53 | 156
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 3 | 2 | 6
  Black/African American | 9 | 7 | 11 | 27
  Caucasian/White | 71 | 70 | 67 | 208
  Multiple | 0 | 1 | 1 | 2
Ethnicity [Number; unit: participants]
  Hispanic/Latino | 5 | 3 | 10 | 18
  Not Hispanic/Latino | 76 | 78 | 71 | 225
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Placebo: N=78, Dysport 500 U: N=80, and Dysport 1000 U: N=80.
  kg/m2 | 26.78 (5.38) | 27.63 (4.61) | 27.58 (5.51) | 27.33 (5.17)
Modified Ashworth Scale (MAS) [Mean (Standard Deviation); unit: units on a scale] — MAS scale is used to assess muscle tone (MT) using a 6-point scale where:0=No increase in MT, 1=Slight increase in MT,1±=Slight increase in MT manifested by a catch followed by minimal resistance throughout remainder of ROM,2=Marked increase in MT through most of ROM but affected part easily moved,3=Considerable increase in MT passive movement difficult or 4=Affected part(s) rigid in flexion or extension. The MAS has been derived for analyses as follows: 0=0 ; 1=1; 1+=2; 2=3; 3=4 and 4=5.
  Placebo:N=79, Dysport 500U:N=80 & Dysport 1000U:N=79.
  units on a scale | 3.9 (0.4) | 3.9 (0.5) | 3.9 (0.4) | 3.9 (0.4)
Disability Assessment Scale (DAS) [Mean (Standard Deviation); unit: units on a scale] — DAS is a 4-point scale used to determine the extent of functional impairment in 4 functional domains (dressing, hygiene, limb position and pain). DAS scale rating: 0=No disability, 1=Mild disability (noticeable but does not interfere significantly with normal activities), 2=Moderate disability (normal activities require increased effort and/or assistance) and 3=Severe disability (normal activities limited). If the subject chose Hygiene as PTT the score collected will be between 0 and 3.
  Placebo: N=79, Dysport 500 U: N=80 and Dysport 1000 U: N=79.
  units on a scale | 2.6 (0.5) | 2.6 (0.5) | 2.5 (0.5) | 2.6 (0.5)

OUTCOME MEASURES:

1. Secondary Outcome: Physician's Global Assessment (PGA) of Treatment Response
Description: PGA is a 9-point scale used to assess global overall treatment response by the investigator (-4: markedly worse, -3: much worse, -2: worse, -1: slightly worse, 0: no change, +1: slightly improved, +2: improved, +3: much improved and +4: markedly improved).
Time Frame: At Week 4
Population: ITT population. Two subjects each from Placebo and Dysport 1000 U had missed PGA assessment at week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dysport 500 U | Dysport 1000 U
Number analyzed (Participants) | 78 | 80 | 78
units on a scale | 0.6 (1.0) | 1.4 (1.1) | 1.8 (1.1)

2. Secondary Outcome: Change From Baseline in DAS Score for the Principal Target of Treatment (PTT)
Description: DAS is a 4-point scale used to determine the extent of functional impairment in 4 functional domains (dressing, hygiene, limb position and pain). DAS scale rating: 0=No disability, 1=Mild disability (noticeable but does not interfere significantly with normal activities), 2=Moderate disability (normal activities require increased effort and/or assistance) and 3=Severe disability (normal activities limited).
  If subject chose 'Hygiene' as PTT the score collected will be between 0 and 3.
Time Frame: From Baseline (Day 1) to Week 4
Population: ITT population. Two subjects each from Placebo and Dysport 1000 U had missed DAS assessment at baseline and week 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dysport 500 U | Dysport 1000 U
Number analyzed (Participants) | 79 | 80 | 79
units on a scale | -0.5 (0.7) | -0.7 (0.8) | -0.7 (0.7)

3. Primary Outcome: Change From Baseline in MAS Score in the Primary Targeted Muscle Group (PTMG)
Description: MAS scale is used to assess muscle tone using a 6-point scale where: 0=No increase in muscle tone, 1=Slight increase in muscle tone manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM) when the part is flexed or extended, 1±Slight increase in muscle tone manifested by a catch followed by minimal resistance throughout the remainder of the ROM, 2=Marked increase in muscle tone through most of the ROM but affected part easily moved, 3=Considerable increase in muscle tone passive movement difficult or 4=Affected part(s) rigid in flexion or extension. The MAS has been derived for analyses as follows: 0=0 ; 1=1; 1+=2; 2=3; 3=4 and 4=5.
Time Frame: From Baseline (Day 1) to Week 4
Population: Intention to treat (ITT) population included all randomized subjects who received at least one injection of study drug and had a MAS score at baseline (pretreatment) and at week 4. Total 5 subjects were excluded from ITT population as they did not have MAS score at baseline or/and at week 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dysport 500 U | Dysport 1000 U
Number analyzed (Participants) | 79 | 80 | 79
units on a scale | -0.3 (0.6) | -1.2 (1.0) | -1.4 (1.1)

ADVERSE EVENTS:
Time Frame: Up to 24±2 weeks
Arm/Group | Placebo | Dysport 500 U | Dysport 1000 U
Serious Adverse Events (participants affected / at risk) | 3/81 | 3/81 | 3/81
Other Adverse Events (participants affected / at risk) | 10/81 | 25/81 | 18/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Dysport 500 U (N=81) | Dysport 1000 U (N=81)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Behcet's syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Dysport 500 U (N=81) | Dysport 1000 U (N=81)
Nasopharyngitis (Infections and infestations) | 1 (1) | 7 (7) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infections (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Gamma glutamyl transferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 2 (2) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No